CLINICAL TRIAL: NCT02584803
Title: Inferior Vena Cava Assessment in Term Pregnancy Using Ultrasound: a Feasibility Study of Subxiphoid and RUQ Views
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 103637
Record Dates: First submitted 2015-10-19; First posted 2015-10-23 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2016-05

CONDITIONS: Hypotension; Hypovolemic Shock
MeSH Terms: conditions — Hypotension; Shock | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Ultrasound — Evaluating the feasibility and efficacy of IVC ultrasound imaging through the RUQ and subxiphoid view in term parturients.
  1. Patient Acceptability of procedure
  2. Patient Comfort:
  3. Ease of exam for the examiner

SUMMARY:
This study is to assess the feasibility of 2 different ultrasound views of the inferior vena cava (IVC), a large vein that returns blood to the heart. Ultrasound is safe in pregnancy and, is regularly used to evaluate the fetus. It is hoped that imaging of the IVC will then allow us to determine the fluid status of the parturient which could be helpful in treating hemodynamic instability. This study will not involve any change in management of the participating patients.

DETAILED DESCRIPTION:
Anesthesiology consultants and trainees with US experience will first perform scans from the RUQ view starting on the mid-axillary line at the T4 intercostal space, looking to obtain a view of the IVC as it enters the right atrium (RA). Following successful acquisition, the examiner will perform scan from the subxiphoid position, looking to obtain the same view of the IVC transitioning into the RA. Primary endpoint will be time to obtaining quality of images. The investigator will use a stopwatch to time acquisition of images. If the duration of scanning exceeds ten minutes, the scan will be discontinued and labeled as failed. Each image will be separately reviewed by 2 different US specialists with extensive US experience. Images will be assessed according to a Likert scale from 1 to 5. (Very poor (1), poor (2), acceptable (3), good (4), very good (5)) Secondary endpoints will be assessed as follows: 1. Acceptability: all patients participating in the study will complete a questionnaire to assess acceptability. 2. Comfort: During the exam the patient will have the option to suspend the scan by stating they are uncomfortable and wish to stop. Each request will be noted and taken into the account at data analysis. Furthermore, patients will be given a questionnaire at the end of the scan and asked to rate their comfort level during procedure according to Likert scale. (Very comfortable (5), comfortable (4), equivocal (3), uncomfortable (2), very uncomfortable (1)) 3. Ease of exam: Examiner will rate the ease of image acquirement according to Likert scale. (impossible (1), difficult (2), equivocal (3), easy (4), very easy (5))

ELIGIBILITY:
Inclusion Criteria:

* Adults pregnant females,
* Age 18-45,
* Term pregnancy Parturients not in established labor Singleton pregnancies

Exclusion Criteria:

* Advanced labor,
* Multiple gestations,
* Maternal or fetal distress,
* BMI > 45.
* Inability to obtain informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Full term pregnant patient coming for elective cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Time to obtaining good Quality IVC images through RUQ and subxiphoid window | 60 seconds

SECONDARY OUTCOMES:
Patient Acceptability of procedure | 10 seconds
  Would you agree to have similar ultrasound scans again?
  Yes/No
patient comfort | 10 seconds
  Please rate your comfort during the ultrasound scan, on a scale of 1 to 5. Where 5 is very comfortable and 0 is not comfortable
Ease of exam for the examiner | 10 seconds
  Ease of exam: Examiner will rate the ease of image acquirement according to Likert scale. (impossible (1), difficult (2), equivocal (3), easy (4), very easy (5)

CONTACTS AND LOCATIONS:
Overall Officials: Indu Singh, Principal Investigator — Western University, Schulish school of Medicine, Department of Anesthesia
Locations (1):
- London Health Science Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dennis A, Arhanghelschi I, Simmons S, Royse C. Prospective observational study of serial cardiac output by transthoracic echocardiography in healthy pregnant women undergoing elective caesarean delivery. Int J Obstet Anesth. 2010 Apr;19(2):142-8. doi: 10.1016/j.ijoa.2009.06.007. Epub 2010 Mar 3. PMID 20202818
- [Result] Dennis AT. Transthoracic echocardiography in obstetric anaesthesia and obstetric critical illness. Int J Obstet Anesth. 2011 Apr;20(2):160-8. doi: 10.1016/j.ijoa.2010.11.007. Epub 2011 Feb 18. PMID 21315578